CLINICAL TRIAL: NCT02934191
Title: Celecoxib for Pain Management After Tonsillectomy
Brief Title: Celecoxib After Tonsillectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-011707
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Results first posted 2019-10-17 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Tonsillectomy
Keywords: Tonsillectomy; Post-operative complications; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Celecoxib; Acetaminophen; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen/Oxycodone + Celecoxib (Experimental): Subjects will take acetaminophen orally (dose 15mg/kg/dose) in scheduled doses every 4 hours for the first 5 days. Subjects will also take celecoxib orally (dose is 6mg/kg twice a day with a maximum dose of 300mg twice a day). The first dose of celecoxib will be given preoperatively, within 1 hour prior to entering the operating room. The second dose will be given at bedtime on the night of surgery and subsequent doses will be given 12 hours apart. Supplemental standard of care oxycodone may be used to control breakthrough pain.
  Interventions: Drug: Celecoxib; Drug: Acetaminophen; Drug: Oxycodone
- Acetaminophen/Oxycodone + Placebo (Active Comparator): Subjects will take acetaminophen orally (dose 15mg/kg/dose) in scheduled doses every 4 hours for the first 5 days. Subjects will also take the placebo orally twice a day. The first dose of placebo will be given preoperatively, within 1 hour prior to entering the operating room. The second dose will be given at bedtime on the night of surgery and subsequent doses will be given 12 hours apart. Supplemental standard of care oxycodone may be used to control breakthrough pain.
  Interventions: Other: Placebo; Drug: Acetaminophen; Drug: Oxycodone

INTERVENTIONS:
Drug: Celecoxib — Dosing will be 6mg/kg twice a day with a maximum dose of 300mg twice a day. All ages will be given the suspension (concentration 100mg/5mL) orally
  Other Names: Celebrex
  Arms: Acetaminophen/Oxycodone + Celecoxib
Other: Placebo — Placebo will have the same appearance, taste and consistency as celecoxib. Placebo will consist of calcium carbonate powder suspended in the same syrup as celecoxib. Dose of elemental calcium is 3 mg/kg/day.
  Other Names: Calcium carbonate placebo
  Arms: Acetaminophen/Oxycodone + Placebo
Drug: Acetaminophen — Acetaminophen syrup at a dose of 15mg/kg/dose will be given every 4 hours for the first 5 days after surgery. After that point, is given as needed.
Drug: Oxycodone — Oxycodone may be used every 4 hours post-operatively to treat breakthrough pain. The most commonly prescribed dose is 0.075mg/kg/dose (suspension) every 4 hours as needed.

SUMMARY:
Tonsillectomy is one of the most common pediatric surgical procedures in the United States. Postoperative pain is substantial, with typical regimens employing narcotic derivatives and acetaminophen for 1-2 weeks after surgery. Recent enthusiasm for use of ibuprofen as an alternative has been tempered by equivocal data on its relative safety in regard to risk of postoperative hemorrhage. The primary objective is to evaluate efficacy of celecoxib for pain control after tonsillectomy in children. The secondary objective is to assess safety in regard to postoperative hemorrhage and adverse events.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial. Subjects will take acetaminophen plus either celecoxib or placebo in regular scheduled doses, and will supplement as needed with standard of care analgesic therapy (oxycodone/acetaminophen).

Celecoxib is approved by the FDA for use in children ages 2 and older for treatment of juvenile rheumatoid arthritis (JRA). Celecoxib is on the Children's Hospital of Philadelphia (CHOP) formulary for use in (1) patients >= 2 years old for JRA, (2) patients >= 12 years old and >=40 kg who have increased risk for gastrointestinal (GI) adverse effects or bleeding concerns precluding use of traditional nonsteroidal anti-inflammatory drugs (NSAIDs), and (3) oncology patients with surface area >= 0.4 square meters for anti-angiogenesis. Celecoxib is approved by the FDA for use in adults for treatment of arthritic conditions, acute/ postoperative pain, and primary dysmenorrhea, and has been widely used since its introduction in 1998.

Setting/Participants:Subjects are healthy children aged 3 to 11 years who undergo tonsillectomy with or without adenoidectomy at any Children's Hospital of Philadelphia (CHOP) location. Subjects with coagulation disorders are excluded. Approximately 300 subjects will be enrolled, 150 in each treatment group.

Study Interventions and Measures: Subjects are provided celecoxib or placebo in scheduled doses every 12 hours for 5 days, then continue until they are pain-free, for a maximum of 10 days. Throughout the study, they are allowed to use oxycodone/acetaminophen as needed for additional pain control, following standard clinical care. Acetaminophen is used around the clock for the first 5 days in all subjects. For 14 days following surgery, subjects record pain levels on validated pain scale instruments, quantity of narcotic medication and acetaminophen required, and time to return to normal diet. All Emergency Department and hospital admissions during the 30 postoperative days are recorded, noting incidence of excess pain, dehydration, hemorrhage, and other complications.

Pain control efficacy is assessed by comparing groups for number of days in which narcotic medication was used, and total quantity of rescue pain medication consumed. Rates of hospital readmission and postoperative hemorrhage, and the need for operative control, are also compared between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 3 to 11 years inclusive.
2. Scheduled to undergo tonsillectomy (with or without adenoidectomy).
3. Weight ≥10 kg.
4. Girls ≥ 11 years of age must have a negative urine/serum pregnancy test on the day of surgery and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
5. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Prior adenotonsillar surgery.
2. Concomitant surgical procedure that adds more than mild additional pain. Note: ear tubes are always permissible.
3. Coagulation disorder, or any other hematologic disorder that affects clotting or results in anemia.
4. Moderate to severe asthma, defined as subjects who either (1) have daily symptoms requiring daily use of short-acting bronchodilators, or (2) had an exacerbation in the last 3 months requiring admission, emergency department (ED) visit, or systemic corticosteroid administration.
5. Any degree of aspirin-sensitive asthma, or any history of asthma exacerbation caused by NSAID use.
6. Severe obstructive sleep apnea, defined as an obstructive apnea-hypopnea index >30 per hour and/or lowest oxygen saturation below 80%
7. Significant chronic pulmonary disease, defined as subjects requiring oxygen therapy, ventilator support, or positive pressure therapy.
8. Significant cardiac disease, defined as any one of the following: cardiovascular disease, structural cardiac anomalies, prior cardiac surgery, or requirement for cardiac anesthesia.
9. Severely obese (weight or body mass index > 95th percentile for age) or underweight (weight <5th percentile for age).
10. History of hepatic or renal disease, or condition that impairs hepatic or renal function.
11. Juvenile rheumatoid arthritis (JRA).
12. History of GI bleeding, or chronic GI condition that would increase risk of bleeding, ulceration, or perforation
13. Hypertension.
14. Craniofacial syndromes.
15. Syndrome or neurologic condition that would hinder accurate assessment of postoperative pain.
16. Inability to feed orally or take oral pain medication.
17. Chronic pain disorders, or otherwise requiring pain medication more than once weekly.
18. Laboratory abnormalities on the preoperative complete blood count (CBC):

    * Hemoglobin < 9 gm/dL
    * Platelet count < 100,000/mm3
19. Any investigational drug use within 30 days prior to enrollment.
20. Pregnant or lactating females.
21. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
22. Hypersensitivity or allergic reactions to celecoxib, aspirin, or other NSAIDs, including asthma flare ups
23. Allergy to sulfonamides or calcium carbonate.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2016-06; Primary Completion 2018-08-17 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Germiller, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giordano T, Durkin A, Simi A, Shannon M, Dailey J, Facey H, Ballester L, Wetmore RF, Germiller JA. High-Dose Celecoxib for Pain After Pediatric Tonsillectomy: A Randomized Controlled Trial. Otolaryngol Head Neck Surg. 2023 Feb;168(2):218-226. doi: 10.1177/01945998221091695. PMID 35412873

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetaminophen/Oxycodone + Celecoxib: Subjects will take acetaminophen orally in scheduled doses every 4 hours for the first 5 days. Subjects will also take celecoxib orally (dose is 6mg/kg twice a day with a maximum dose of 300mg twice a day). The first dose of celecoxib will be given preoperatively, within 1 hour prior to entering the operating room. The second dose will be given at bedtime on the night of surgery and subsequent doses will be given 12 hours apart. Supplemental standard of care oxycodone may be used to control breakthrough pain.
  Celecoxib: Dosing will be 6mg/kg twice a day with a maximum dose of 300mg twice a day. All ages will be given the suspension (concentration 100mg/5mL) orally.
- Acetaminophen/Oxycodone + Placebo: Subjects will take acetaminophen orally in scheduled doses every 4 hours for the first 5 days. Subjects will also take the placebo orally twice a day. The first dose of placebo will be given preoperatively, within 1 hour prior to entering the operating room. The second dose will be given at bedtime on the night of surgery and subsequent doses will be given 12 hours apart. Supplemental standard of care oxycodone may be used to control breakthrough pain.
  Placebo: Placebo will have the same appearance, taste and consistency as celecoxib. Placebo will consist of calcium carbonate powder suspended in the same syrup as celecoxib. Dose of elemental calcium is 3 mg/kg/day.
Period: Overall Study
Arm/Group | Acetaminophen/Oxycodone + Celecoxib | Acetaminophen/Oxycodone + Placebo
Started | 87 | 85
Completed | 87 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen/Oxycodone + Celecoxib | Acetaminophen/Oxycodone + Placebo | Total
Number analyzed (Participants) | 87 | 85 | 172
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6.27 [4.74 to 7.75] | 5.72 [4.44 to 6.96] | 6.03 [4.48 to 7.37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 46 | 95
  Male | 38 | 39 | 77
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87 | 85 | 172

OUTCOME MEASURES:

1. Primary Outcome: Difference in Number of Days Requiring Rescue Pain Medication
Description: The number of days on narcotic pain medication following surgery will be compared between the two treatment groups
Time Frame: 2 weeks post-operative
Population: Subjects with evaluable data
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Acetaminophen/Oxycodone + Celecoxib | Acetaminophen/Oxycodone + Placebo
Number analyzed (Participants) | 73 | 67
Days | 5.00 (3.35) | 5.75 (3.82)

2. Primary Outcome: Difference in Amount of Rescue Pain Medication Consumed
Description: The total amount of rescue pain medication consumed in the 2-week postop period will be compared between the two treatment groups.
Time Frame: 2 weeks post-operative
Population: Subjects with evaluable data
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Acetaminophen/Oxycodone + Celecoxib | Acetaminophen/Oxycodone + Placebo
Number analyzed (Participants) | 73 | 67
mg/kg | 1.03 (1.12) | 1.40 (1.45)

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events were collected for the 30 day postoperative period, and were collected systematically from the day 3, day 14, day 30 telephone calls, and the Study Diary
Arm/Group | Acetaminophen/Oxycodone + Celecoxib | Acetaminophen/Oxycodone + Placebo
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/85
Serious Adverse Events (participants affected / at risk) | 9/87 | 7/85
Other Adverse Events (participants affected / at risk) | 78/87 | 50/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen/Oxycodone + Celecoxib (N=87) | Acetaminophen/Oxycodone + Placebo (N=85)
Hemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 6 (6) — Surgical site hemorrhage
Dehydration (General disorders) | 4 (4) | 1 (1) — Dehydration resulting in admission
Dental infection (Infections and infestations) | 1 (1) | 0 (0) — Dental infection with facial swelling
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Gastroenteritis with admission
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen/Oxycodone + Celecoxib (N=87) | Acetaminophen/Oxycodone + Placebo (N=85)
Nausea / Vomiting (Gastrointestinal disorders) | 19 (19) | 10 (10)
Abdominal Pain (Gastrointestinal disorders) | 31 (31) | 26 (26)
constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 3 (3)
Headache (General disorders) | 11 (11) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT02934191/Prot_SAP_000.pdf